CLINICAL TRIAL: NCT00996684
Title: Resolution of Vitreomacular Adhesion (VMA) Associated With Neovascular Age Related Macular Degeneration (AMD) With Intravitreal Microplasmin
Brief Title: Study of Intravitreal Microplasmin in Relieving Vitreo-Macular Adhesion in Neovascular Age-related Macular Degeneration
Acronym: AMD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: ThromboGenics (Industry)
Responsible Party: Principal Investigator, Steven Schwartz, Chief, Retina Division, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JSEI-TG-AMD-001
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Macular Degeneration
Keywords: Wet age related macular degeneration (AMD); Wet AMD; Vitreomacular adhesion (VMA); Vitreomacular traction (VMT); Neovascular age related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — microplasmin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- microplasmin, intravitreal injection (Experimental): Subjects will receive one intravitreal injection of microplasmin on Day 0.
  Interventions: Drug: Microplasmin
- Placebo (Placebo Comparator): Subjects will receive one intravitreal injection of the placebo on Day 0.
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: Microplasmin — Microplasmin, 1.875 mg, will be given by intravitreal injection,on Day 0.
  Arms: microplasmin, intravitreal injection
Drug: Placebo control — The placebo control will be the microplasmin vehicle without the microplasmin.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether microplasmin given by intravitreal injection is effective and safe for the treatment of wet age-related macular degeneration (AMD) in patients who have focal vitreomacular adhesion (VMA)

DETAILED DESCRIPTION:
The human vitreous gel undergoes progressive liquefaction with age. Concurrent with the process of vitreous liquefaction, there is a weakening of the adhesion at the vitreoretinal interface between the cortical vitreous gel and the inner limiting lamina. Posterior vitreous detachment (PVD) is a separation of the cortical vitreous get from the inner limiting lamina. PVD is usually a sudden event during which liquefied vitreous from the center of the vitreous body bursts through a hole in the posterior vitreous cortex and then dissects the residual cortex gel away from the inner limiting lamina. If there is residual vitreoretinal traction around the break, this process may induce a tear in the retina that can in turn result in rhegmatogenous retinal detachment, macular hole, or cystoid macular edema. The importance of the vitreous in the progression of diabetic retinopathy may also extend beyond tractional considerations. For example, it is believed that the vitreous serves as scaffolding for new vessel formation and may also contribute to molecular imbalances that lead to retinopathy progression. Therefore, total PVD, by releasing vitreoretinal traction as well as other potential mechanisms, may be beneficial in various vitreoretinal diseases such as neovascular AMD.

Vitreomacular adhesion (VMA) in exudative (wet) AMD may be associated with poor prognosis in patients with AMD. This trial is primarily aimed at showing that release of VMA can be induced by microplasmin, a proteolytic enzyme, in patients with wet AMD, and that microplasmin is safe in patients w/ neovascular (wet) AMD. Secondary endpoint will be assessment of improved AMD outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 50 years or older
* Presence of focal vitreomacular adhesion as seen by OCT
* BCVA of 20/800 or better in non-study eye
* Presence of active choroidal neovascular membrane
* Written informed consent obtained from subject prior to inclusion in the trial

Exclusion Criteria:

* Subjects who have previously received microplasmin
* Subjects with any vitreous hemorrhage or any other vitreous opacification which precludes adequate examination or investigation of study eye
* Patient with uncontrolled glaucoma including IOP >25 mm Hg
* Subjects who have had vitrectomy or retinal detachment or who are aphakic or highly myopic (>8.0 D) in the study eye
* Subjects who are pregnant or of child-bearing potential not utilizing an acceptable form of contraception. Acceptable methods include intrauterine device, oral, implanted or injected contraceptives, and barrier methods with spermicide.
* Subjects who, in the Investigator's view, will not complete all visits and investigations
* Patient who have PDT or any intravitreal injection in the last 10 days. Patients who in the examiners opinion will need intravitreal injection in the next 10 days (apart from microplasmin).
* Patients who have participated in an investigational drug trial in the past 30 days.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the proportion of patients in whom there is release of vitreomacular traction as assessed by ultrasonography, optical coherence tomography and physical examination | Day 28

SECONDARY OUTCOMES:
Total number of ranibizumab injections following microplasmin in those with PVD compared with those without PVD | 12 months
Change in mean macular thickness | Day 28 and month 12
Mean change in ETDRS visual acuity | Day 28 and Month 12
Incidence and severity of ocular adverse events | Day 28 and Month 12
Incidence and severity of nonocular adverse events | Day 28 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Schwartz, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Jules Stein Eye Institute/UCLA, Los Angeles, California, United States